CLINICAL TRIAL: NCT03933852
Title: Observational Study on Chronic Myeloid Leukemia Patients in Any Phase Treated With Ponatinib (Iclusig®) at Any Dose
Acronym: Ponderosa
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Andreas Hochhaus, Director Clinic of Internal Medicine II, University of Jena
Other Study IDs: Ponderosa
Record Dates: First submitted 2019-04-08; First posted 2019-05-01 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Chronic Myeloid Leukemia, Chronic Phase
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Additional information is needed to characterize the safety profile of ponatinib as it is used in routine clinical practice in Europe. This observational cohort study will provide a real-life picture of ponatinib use in clinical practice and additional quantification and characterization of adverse events (AEs) and their outcomes in patients with Chronic Myeloid Leukemia in any phase treated with ponatinib.

DETAILED DESCRIPTION:
This study is a multicentre, long-term, prospective and retrospective, observational cohort study of patients who are treated with ponatinib. The study is non-interventional; all Treatment decisions are made at the discretion of the patient's healthcare provider (HCP) and are not mandated by the study design or protocol.

A heterogeneous sample of oncology practice sites in Germany (both Hospitals and Field based Haematologists) treating adult patients with Chronic Myeloid Leukemia in any phase using ponatinib will be selected for participation in the study. Eligible, consenting patients initiating treatment with ponatinib will be enrolled into the prospective part of the study. Eligible consenting patients with Chronic Myeloid Leukemia in any Phase that have initiated ponatinib outside clinical trial after its approval in Germany will be enrolled in the retrospective part of the study.

Approximately 100 patients will be enrolled from approximately 50 sites. The patient enrolment period is estimated to be approximately two years. Patients who experience an Adverse Event (AE) during treatment or within the 30 days post discontinuation will be followed for 12 months to determine the consequences of the Adverse Event. Data on patient's history, patient's data at baseline, ponatinib treatment, Adverse Events, all medications received, and efficacy measures will be collected during the study in conjunction with routine care visits, anticipated to be approximately every 3 months.

Information on any new therapies, including treatment for Chronic Myeloid Leukemia and other medications will be collected during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥18 years) with Chronic Myeloid Leukemia in any phase who are initiating ponatinib monotherapy, or for whom ponatinib monotherapy was initiated after ponatinib approval in Germany. [The decision to prescribe ponatinib must have been made prior to enrolment in the study. Patients enrolled in the retrospective part of the study may or may not be still on ponatinib treatment at the time informed consent is given. These retrospective patients should have started Treatment after 02.02.2015.].
* Patients who have the ability to understand the requirements of the study, and provide written informed consent to comply with the study data collection procedures.
* Patients with a minimum life expectancy of 3 months

Exclusion Criteria:

* Patients previously treated with investigational ponatinib (within a clinical trial)
* Patients receiving an investigational agent
* Patients who are pregnant and/or breastfeeding
* Patients who are pregnant and/or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients with Chronic Myeloid Leukemia in any phase that are initiating or have initiated treatment with ponatinib and who meet the enrolment criteria and provide informed consent. A group of patients, for whom the decision of starting ponatinib has already been made, but in whom ponatinib has not yet been started, will be identified prospectively and invited to enrol into the study. The study enrolment date is the date the informed consent is signed. An additional group of patients who have received or are receiving ponatinib treatment outside clinical trials will be invited to join the retrospective part of the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-07-08 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Cytogenetic response | through study completion, an average of 3 years
  Achievement of cytogenetic Response (percentage of Ph+ metaphases)
Molecular response | through study completion, an average of 3 year
  BCR-ABL in % (lower is better)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Hochhaus, Principal Investigator — University Hospital Jena
Locations (1):
- University Hospital Jena, Jena, Germany

IPD SHARING:
Plan to Share IPD: No